CLINICAL TRIAL: NCT01694316
Title: Use of a Novel Neuroplasticity-based Neurobehavioral Intervention for PTSD - A Nationwide, Online Study
Brief Title: Use of a Novel Neuroplasticity-based Neurobehavioral Intervention for PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Amit Etkin, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-24890
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Anxiety; Depression
Keywords: Computerized neurobehavioral intervention
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Engaging in Computerized tasks (Active Comparator): Participants will log into a personalized website and engage in computerized tasks online.
  Interventions: Behavioral: Computerized Neurobehavioral Intervention
- Neurobehavioral computerized tasks (Experimental): Participants will log into a personalized website and engage in computerized tasks online.
  Interventions: Behavioral: Computerized Neurobehavioral Intervention

INTERVENTIONS:
Behavioral: Computerized Neurobehavioral Intervention — Targeted, computerized interventions completed from the participants' own home on a computer.

SUMMARY:
The present study will explore the effectiveness of a computer based neurobehavioral intervention in alleviating symptoms and improving emotion regulation in individuals with PTSD. It will increase understanding of psychopathology at a neural-circuit level and aid development of new non-pharmacological treatment for PTSD. The study is managed by the Etkin Lab at Stanford University in California, but participants from the entire US are welcome to participate as the study is delivered online.

ELIGIBILITY:
Inclusion Criteria:

* current PTSD
* internet access

Exclusion Criteria:

* lifetime psychotic disorder,
* past-year substance dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
WebNeuro Computerized Cognitive and Affective Assessment Battery | Baseline and 3-month
  Age and gender-normed Z scores for the following measures:
  Sustained attention accuracy, Sustained attention lapses, Sustained attention false alarms, Working memory capacity, Visual scanning speed, Inhibition executive control, Processing speed, Maze completion executive control accuracy, Maze completion executive control speed, Immediate verbal memory, Delayed verbal memory, Inhibitory motor control accuracy, Inhibitory motor control lapses, Facial affect identification accuracy (happy, fearful, angry, sad, and disgusted), Facial affect identification speed (happy, angry, fearful, sad, or disgusted), Facial affect identity recognition accuracy (happy, angry, sad, fearful, or disgusted), Facial affect identity recognition speed (happy, sad, angry, fearful, or disgusted), Emotional conflict reaction time slowdown, Regulation of emotional conflict reaction time slowdown

SECONDARY OUTCOMES:
Clinician-assessed PTSD symptoms | Baseline and 3-month
  Total and symptom sub scale scores from the Clinician-Administered PTSD Scale for DSM-IV (CAPS)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Department of Psychiatry and Behavioral Sciences, Stanford, California, United States

REFERENCES:
- [Derived] Fonzo GA, Fine NB, Wright RN, Achituv M, Zaiko YV, Merin O, Shalev AY, Etkin A. Internet-delivered computerized cognitive & affective remediation training for the treatment of acute and chronic posttraumatic stress disorder: Two randomized clinical trials. J Psychiatr Res. 2019 Aug;115:82-89. doi: 10.1016/j.jpsychires.2019.05.007. Epub 2019 May 8. PMID 31125916
- See also: Related Info — https://sites.google.com/site/veteranonlinestudy/